CLINICAL TRIAL: NCT04702438
Title: SMART Family-Link Project: Zentangle to Promote Family Well-being in Hong Kong
Brief Title: Zentangle to Promote Family Well-being in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UW 19-489-1
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-01

CONDITIONS: Family Research
Keywords: Family Well-being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ICT activities — Family interventions using ICT to promote family communication, sharing happiness with family members, and well-being in the community.

SUMMARY:
In the past few decades, Information and Communications Technology (ICT) have rapidly developed as effective, and probably the most cost-effective tools to connect most aspects of family lives. Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also an increasing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

To gain more understanding of the potential new avenues of using ICT in programme implementation, The Hong Kong Jockey Club Charities Trust has initiated the Jockey Club SMART Family-Link Project in collaboration with The University of Hong Kong (HKU) and non-governmental organizations (NGOs). This project aimed at helping 26 NGO-operated Integrated Family Service Centres and Integrated Service Centres (Centres), making effective use of information and communications technology (ICT) and data analytics, to enhance the quality and efficiency of their family service. The present study aims to supplement the existing services and interventions delivered by the FRU, FSU and FCU, a series of brief ICT-based family interventions that promote family communication, cohesion, support and well-being and improve the efficiency and effectiveness of ICT-based interventions.

DETAILED DESCRIPTION:
With the increasing use of ICT, family information can be easily accessed. According to the findings from FHinTs 2016, ICT was increasingly used as a method of family information seeking: 66.7% of respondents sought family information from online websites, compared with 53.6% in 2009. About 30.9% sought family information from social media such as Facebook, and 22.8% sought family information from instant messaging platforms such as WhatsApp. Family information such as recreation (46.6%), family health (22.9%) and elderly-related topics (17.9%) was most commonly sought. Also, family information seeking was associated with higher levels of family health, happiness, harmony, and overall family well-being. The associations were observed regardless of the type of sharing methods, such as face-to-face sharing or sharing via ICT means.

Alongside the growth in popularity of ICTs and its role in promoting family well-being, there is also a growing appreciation that ICTs such as internet-enabled devices and web-based applications can offer many advantages compared to traditional face-to-face approaches when delivering behaviour change programmes.

Family services in Hong Kong In light of the review on family services in Hong Kong in 2000, pilot projects on the Integrated Family Service Centre (IFSC) service mode were conducted in 2002. Having received positive feedback from the community on the pilot projects, 61 IFSCs were established in 2004 to provide public-funded family services in Hong Kong. These IFSCs comprise three important components, including the family resource unit (FRU), family support unit (FSU), and family counselling unit (FCU) to provide preventive, supportive, and remedial services respectively. They are operated by the Social Welfare Department and subvented non-governmental organizations to support and strengthen individuals and families, particularly single parents, new arrivals, ethnic minorities, and deprived families receiving Comprehensive Social Security Assistance (CSSA), in the community.

Jockey Club SMART Family-Link Project Family well-being is the cornerstone of a harmonious society, and early support for families in need will avert a crisis. The Hong Kong Jockey Club Charities Trust has funded to a four-year (2018-2021) "Jockey Club SMART Family-Link Project" to advance the use of Information and Communications Technology ("ICT") in family services. Interventions leveraging ICT (i-Action) is one of the project components, which leverage ICT to help social workers offer ICT-based interventions in their work to add to their face-to-face interventions. ICT tools and mobile apps will be designed and interactive games will be provided to engage children and young family service users through e-platforms. Social workers will also be able to connect with service users between face-to-face sessions using these e-platforms.

The present study aims to reduce stress, enhance resilience and promote personal and family well-being through Zentangle. We will conduct quantitative and qualitative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Family service users
* Chinese-speaking
* Aged 18 years and above
* Able to complete the questionnaire

Exclusion Criteria:

* Subjects who fail to meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Social service users
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction to the Zentangle programme | Immediately after the activities
  Outcome-based questions will be used to assess the level of satisfaction toward the general performance of the community activities. The score for each question ranges from 1 to 5. Higher scores indicate higher satisfaction.

SECONDARY OUTCOMES:
Change in Family communication | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess the communication with family members. The score for each question ranges from 0 to 10. Higher scores indicate better family communication.
Change in Family relationship | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess the relationship with family members. The score for each question ranges from 0 to 10. Higher scores indicate better family relationship.
Change in Family support and care | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess the family support and care. The score for question ranges from 0 to 10. Higher scores indicate more family support and care.
Change in Resilience | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess resilience. The score for question ranges from 0 to 10. Higher scores indicate higher resilience.
Change in Healthy living habits | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess healthy living. The score for question ranges from 0 to 10. Higher scores indicate healthier living.
Change in Personal happiness | Baseline, 1-month and 2-month follow up
  Outcome based question will be used to assess personal happiness. The score for question ranges from 0 to 10. Higher scores indicate more personal happiness.
Change in Stress level | Baseline, 1-month and 2-month follow up
  Change assessed by the Perceived Stress Scale (PSS). A higher score means a worse outcome.
Change in Negative emotions | Baseline, 1-month and 2-month follow up
  Change assessed by the Patient Health Questionnaire-4. A higher score means a worse outcome.
Change in Family well-being | Baseline, 1-month and 2-month follow up
  Change assessed by a 3-item Family well-being scale. A higher score means a better outcome.
Change in Self-efficacy in managing stress | Baseline, 1-month and 2-month follow up
  Outcome-based questions will be used to assess self-efficacy in managing stress. Higher score indicates higher self-efficacy.
Change in Knowledge and attitudes towards and practice of Zentangle | Baseline, 1-month and 2-month follow up
  Change assessed by outcome-based questions. A score of each question ranges from 1-5. A higher score a better outcome.
Perceived benefits of Zentangle | 1-month and 2-month follow up
  Assessed by outcome-based questions with categorical choices

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong Island, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breitenstein SM, Gross D, Christophersen R. Digital delivery methods of parenting training interventions: a systematic review. Worldviews Evid Based Nurs. 2014 Jun;11(3):168-76. doi: 10.1111/wvn.12040. Epub 2014 May 19. PMID 24842341
- [Background] Enebrink P, Hogstrom J, Forster M, Ghaderi A. Internet-based parent management training: a randomized controlled study. Behav Res Ther. 2012 Apr;50(4):240-9. doi: 10.1016/j.brat.2012.01.006. Epub 2012 Jan 30. PMID 22398153
- [Background] Gross D, Johnson T, Ridge A, Garvey C, Julion W, Treysman AB, Breitenstein S, Fogg L. Cost-effectiveness of childcare discounts on parent participation in preventive parent training in low-income communities. J Prim Prev. 2011 Dec;32(5-6):283-98. doi: 10.1007/s10935-011-0255-7. PMID 22134677
- [Background] Kingston D, Janes-Kelley S, Tyrrell J, Clark L, Hamza D, Holmes P, Parkes C, Moyo N, McDonald S, Austin MP. An integrated web-based mental health intervention of assessment-referral-care to reduce stress, anxiety, and depression in hospitalized pregnant women with medically high-risk pregnancies: a feasibility study protocol of hospital-based implementation. JMIR Res Protoc. 2015 Jan 16;4(1):e9. doi: 10.2196/resprot.4037. PMID 25595167
- [Background] Bert SC, Farris JR, Borkowski JG. Parent training: implementation strategies for adventures in parenting. J Prim Prev. 2008 May;29(3):243-61. doi: 10.1007/s10935-008-0135-y. PMID 18446440
- [Background] Treisman GJ, Jayaram G, Margolis RL, Pearlson GD, Schmidt CW, Mihelish GL, Kennedy A, Howson A, Rasulnia M, Misiuta IE. Perspectives on the Use of eHealth in the Management of Patients With Schizophrenia. J Nerv Ment Dis. 2016 Aug;204(8):620-9. doi: 10.1097/NMD.0000000000000471. PMID 26828911
- [Background] Proudfoot J. The future is in our hands: the role of mobile phones in the prevention and management of mental disorders. Aust N Z J Psychiatry. 2013 Feb;47(2):111-3. doi: 10.1177/0004867412471441. No abstract available. PMID 23382507